CLINICAL TRIAL: NCT04581720
Title: Determination of the Minimum Current for Train-of-four Monitoring by Acceleromyography and Electromyography During the Recovery From General Anesthesia
Brief Title: Minimum Current for Train-of-four Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Sooyoung Cho, Clinical Assistant Professor, Ewha Womans University Mokdong Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-06-017
Record Dates: First submitted 2020-09-27; First posted 2020-10-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Anesthesia; Anesthesia Recovery Period; Neuromuscular Blockade
MeSH Terms: interventions — Neuromuscular Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): The participants will be applied AMG and EMG on each arm of both arms when they finish routine monitoring before the induction of general anesthesia. After the participants being unconscious, we will find each participant's supramaximal current before injecting the neuromuscular blocking agents. During the operation, when the TOF count reaches 4 again and the height of T1 reaches 50% of baseline, we perform TOF tests using 4 currents (Supramaximal current, 0.7×supramaximal current, 0.5×supramaximal current, 0.3×supramaximal current), three times for respective current to figure out that low current can show the same level of TOF ratio as the supramaximal current. When the operation ends and the T1 reaches 100% of baseline, we perform TOF tests with 4 currents again. In the postanesthesia care unit, we use EMG only and perform TOF tests with 4 currents again. The participants can feel pain by the stimulants during the tests, so if they refuse the tests, we stop the tests and record it.
  Interventions: Device: Train-of-four (TOF)

INTERVENTIONS:
Device: Train-of-four (TOF) — Give 4 electrical stimulants on the ulnar nerve to see if the 4 responses (T1 ~ T4) of adductor pollicis fade or not. If there's no neuromuscular block, it shows no fade, or it fades. When an operation is over under general anesthesia, we use the ratio of the height of T4 to T1, and the ratio is over 90%, the neuromuscular block is recovered enough to extubation.

SUMMARY:
Neuromuscular monitoring during general anesthesia is important to make sure adequate muscle relaxation during operation and adequate recovery of muscle power and spontaneous breathing during emergence from general anesthesia. The neuromuscular monitoring is usually using electrical stimulants and the method called train-of-four (TOF) is representative. Because it uses electrical stimulants, the patients could be uncomfortable and feel pain during the monitoring when the patients are conscious. Lowering the current of the stimulants would be helpful in reducing the pain, but there is a concern that the TOF results performed in lower current would be underestimated or inaccurate. Therefore, the investigators want to find the minimal current for TOF monitoring that shows adequate TOF results.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65
* Scheduled for an elective surgery
* ASA physical status 1 or 2

Exclusion Criteria:

* BMI > 25 kg/m2
* Neuromuscular disease
* Decreased renal function
* Neurologic disorder
* Impossible to cooperate or communicate

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Minimal current for TOF | During the operation, from the height of T1 reaches back to the baseline, to the extubation of tracheal tube when the general anesthesia is over.
  The minimal current among the four currents we use which is showing not significantly lower TOF ratio than TOF ratio of supramaximal stimulant.

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea